CLINICAL TRIAL: NCT01829581
Title: German-wide Multicenter Analysis of Oral Anticoagulant-associated Intracerebral Hemorrhage
Brief Title: geRman-widE mulTicenter Analysis of oRal Anticoagulation-associated intraCerebral hEmorrhage
Acronym: RETRACE
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: Multicenter Analysis OAC-ICH
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: OAC-ICH; Acute Management of OAC-ICH; Resumption of OAC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- oral anticoagulation associated intracerebral hemorrhage
  Interventions: Other: no intervention, only descriptive data analysis

INTERVENTIONS:
Other: no intervention, only descriptive data analysis

SUMMARY:
Intracerebral hemorrhage [ICH] is the most feared complication of anticoagulant therapy [OAC]. Evidence regarding acute therapeutic interventions as well as secondary treatment approaches is still limited. Therefore, this German-wide observational cohort study will retrospectively identify and evaluate all OAC-associated ICH patients that have been admitted to the 20 participating tertiary centres over a 5-year period. The main focus of this investigation, besides epidemiological aspects, will be the (i) acute management of OAC-ICH, (ii) secondary therapy (anticoagulant management) and (iii) long-term outcome after OAC-ICH.

DETAILED DESCRIPTION:
Stroke in general is one of the leading causes for death and disability in the industrialized world. Cardiac thromboembolisms are a major contributor to ischemic infarction and the most frequent reason is atrial fibrillation [afib]. The prevalence of afib is constantly increasing within the ageing population and its established therapy (oral anticoagulation) increases alongside. Therefore, rates of OAC-ICH are expected to increase simultaneously. As compared to spontaneous ICH, OAC-ICH is associated with larger ICH-volumes, an increased mortality and poorer functional outcome. Nevertheless, only limited evidence is available for the treatment of such severely injured patients. The only sound benefit is reported for the strategy of "INR-reversal as soon as possible". More detailed therapeutic approaches and guidelines are not well established. Many questions regarding the acute treatment strategy remain to be investigated (modus of INR reversal, prevention of hematoma growth, operative procedures, aso).

Moreover, the most pressing questions that need to be answered relate to coagulation management after OAC-ICH. Would patients benefit from resumption of OAC? Which patients would benefit and when? What are the complication rates (thromboembolic versus bleedings) according to which treatment? How is outcome influenced by the different therapeutic strategies?

This observational cohort study will try to strengthen the therapeutic evidence for OAC-ICH treatment by retrospective data-pooling of 20 nation-wide tertiary hospitals in Germany. Patients will be identified from medical records by the diagnosis of ICH and concomitantly present intake OAC (INR>1.4) during a time period from 2006-2010. Only patients with ICH associated to OAC will be included, other secondary cause i.e. tumors, trauma, vascular malformations etc. will be excluded.

Following parameters will be evaluated: + prior medical history (CHADS-VASC-Score, HAS-Bled Score, risk factors) functional status prior admission; + Timing of symptoms until - admission, - imaging, - therapy initiation; + acute therapy (INR reversal, blood pressure, hematoma growth); + complications and treatment (thrombosis-prophylaxis, infections, transfusions, etc.); + Mortality rates (discharge, 3 months and 1 year, overall long-term); + functional outcome mRS (discharge, 3 months and 1 year, overall long-term); + secondary prophylaxis (OAC vs. platelet inhibitors); + bleedings versus thromboembolic-events.

ELIGIBILITY:
Inclusion Criteria:

* between 2006-2010 in one of the participating centers hospitalized patients with OAC-ICH

Exclusion Criteria:

* secondary ICH other than OAC-ICH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with oral anticoagulation (INR>1.4) associated intracerebral hemorrhage
Sampling Method: Probability Sample
Enrollment: 1205 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Long-term functional outcome | 1 year
  * In-hospital mortality
  * Functional status at discharge
  * Functional short-term outcome (modified Rankin Scale at 3 months)
  * Functional long-term outcome (modified Rankin Scale at 12 months)
Secondary prophylaxis and occurrence of ischemic vs hemorrhagic events | 1 year
Modus of INR reversal | 72 hours
  agent used for INR reversal; timing of INR normalization; occurrence of hemorrhage growth?

CONTACTS AND LOCATIONS:
Overall Officials: Hagen B. Huttner, MD, Principal Investigator — Department of Neurology, University of Erlangen-Nuremberg, Germany

REFERENCES:
- [Derived] Kuramatsu JB, Gerner ST, Schellinger PD, Glahn J, Endres M, Sobesky J, Flechsenhar J, Neugebauer H, Juttler E, Grau A, Palm F, Rother J, Michels P, Hamann GF, Huwel J, Hagemann G, Barber B, Terborg C, Trostdorf F, Bazner H, Roth A, Wohrle J, Keller M, Schwarz M, Reimann G, Volkmann J, Mullges W, Kraft P, Classen J, Hobohm C, Horn M, Milewski A, Reichmann H, Schneider H, Schimmel E, Fink GR, Dohmen C, Stetefeld H, Witte O, Gunther A, Neumann-Haefelin T, Racs AE, Nueckel M, Erbguth F, Kloska SP, Dorfler A, Kohrmann M, Schwab S, Huttner HB. Anticoagulant reversal, blood pressure levels, and anticoagulant resumption in patients with anticoagulation-related intracerebral hemorrhage. JAMA. 2015 Feb 24;313(8):824-36. doi: 10.1001/jama.2015.0846. PMID 25710659